CLINICAL TRIAL: NCT03989323
Title: A Clinical and Biological Prospective Database of Patients Treated With Anticancer Immunotherapy and Follow up of Their Immune-related Adverse Events irAE
Acronym: IMMUCARE-BASE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0816
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples (36 mL) will be collected at the time of the first and second immunotherapy administrations, during routine care. In the case of grade 3 or 4 toxicities, blood samples will be collected as well at the time of irAE onset.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with immunotherapy: Patients receiving for the first time an immunotherapy treatment for their cancer (Checkpoints inhibitors, such as PD-1 or PD-L1 or CTLA4…). Patients will be enrolled before starting the immunotherapy treatment and will be followed up for 5 years or until the permanent discontinuation of the immunotherapy treatment to describe the arm.
  Interventions: Other: Estimation of the incidence of the irAE

INTERVENTIONS:
Other: Estimation of the incidence of the irAE — Assessment of the incidence of the irAE in patients treated with immunotherapy at the Hospices Civils de Lyon (irAE of all grades and from all organs) and creation of a biological collection of blood, plasma, serum and PBMCs from patients before treatment, under treatment and at the onset of irAEs.

SUMMARY:
The number of patients affected by cancer and treated with immunotherapy is continuously increasing. With the advent of these new therapies, the investigators observe the emergence of new and unexpected toxicities. The care of patients treated with these molecules require the development of multidisciplinary skills and the introduction of a professional network capable of taking care of immunotherapy related toxicity (irAE) that can affect different organs and for which immediate and effective interventions are necessary for patient survival.

IMMUCARE-BASE will comprehensively enable the collection, of clinical and biological data of patients treated with anticancer immunotherapy. The creation of this database is essential to identify clinico-biological factors predisposing to toxicity, and to define the best strategies to prevent the early onset of irAE and/or to treat them. Ultimately, the objective of this database is to collect enough data to be able to personalise in the future the immunotherapy treatment according to the benefits and to anticipate risks for each patient.

The objective of the biological collection is to perform ancillary studies for understanding mechanism leading to toxicity and for the development of research programs in the field of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patient starting anticancer immunotherapy treatment(immune checkpoint inhibitors like anti-PD-1, anti-PD-L1, anti-CTLA4, anti-Lag-3, anti-Tim-3, anti-TIGIT or other new anticancer immunotherapy) in monotherapy or associatied with other anticancer molecules.
* Patient who had already received immunotherapy can be eligible to IMMUCARE-BASE provided that the last immunotherapy treatment had been administered > 6 months ago.
* Patient who received written information about IMMUCARE-BASE.
* Patient receiving immunotherapy as a part of a clinical trial can be eligible to IMMUCARE-BASE according to the indications given by the promoter of this trial.
* Patient in a clinical trial which includes a combination of therapy with one of the drugs administered in a blind manner vs placebo, can be eligible to IMMUCARE-BASE provided that (i) the treatment administered in a blind manner is not the immunotherapy and (ii) the clinical trial allows concomitant participation of a patient in another non-interventional study.
* A Patient that has been already included in IMMUCARE-BASE and who terminates the study because of a change of treatment, can be included again in IMMUCARE-BASE if he/she agrees and provided that (i) is the new treatment includes immunotherapy (alone or in association with other anticancer molecules) and (iii) the new immunotherapy treatment is administered after 6 months from the last administration of the previous immunotherapy.

Inclusion criteria specific to the biological collection:

-Signature of the informed consent.

Exclusion Criteria:

* Patient who had received immunotherapy within 6 months before entering in IMMUCARE-BASE
* Minor patient
* Pregnant women
* Patient under juridical protection
* Patient refusal to participate.

Exclusion criteria for the biological collection:

* Weight ≤ 50kg
* Haemoglobin < 90g/L at the time of the inclusion
* Patient participating in clinical trials where blood samples are taken for ancillary studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer and starting anticancer immunotherapy (-immune checkpoint inhibitors: anti-PD-1, anti-PD-L1, anti-CTLA4, anti-Lag-3, anti-Tim-3, anti-TIGIT or other new emerging immune checkpoint inhibitors).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Estimation of the incidence of immunotherapy-related toxicities (all grades, of all organs, in real life) in patients treated for the first time with anticancer immunotherapy and enrolled in the "IMMUCARE-BASE" clinical database | 10 years
  Patients can be treated with immunotherapy alone, or in association with other immunotherapies, or association with chemotherapies, targeted therapies or radiotherapy. It will include all types of cancers that can be treated with immunotherapy, also including patients that are in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan LOPEZ, MD, Study Director — Hospices Civils de Lyon
Locations (5):
- France (5):
  - Hôpital L. Pradel, Bron
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital E Herriot, Lyon
  - Centre Hospitalier LYON SUD, Pierre-Bénite